CLINICAL TRIAL: NCT06019975
Title: FDG-PET in the Diagnosis of Autoimmune Encephalitis
Acronym: PEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: PEA
Record Dates: First submitted 2023-08-04; First posted 2023-08-31 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Autoimmune Encephalitis
Keywords: Autoimmune Encephalitis; FDG-PET; SPM
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune Encephalitis patients: Patients with autoimmune encephalitis admitted to the centers, who underwent a brain FDG-PET during the course of their disease trajectory.
  Interventions: Diagnostic Test: FDG-PET

INTERVENTIONS:
Diagnostic Test: FDG-PET — Brain FDG-PET

SUMMARY:
The goal of this retrospective observational study is to compare brain fluorodeoxyglucose-positron emission tomography (FDG-PET) of patients with autoimmune encephalitis, normal controls and patients with Alzheimer's disease (AD). The main question it aims to answer is:

•is there a specific pattern of brain metabolism in patients with autoimmune encephalitis Participants data and images will be retrospectively collected from hospital records, and FDG-PET images will be analyzed by means of statistical parametric mapping (SPM). Controls will be selected from validated public databases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune encephalitis according to clinical criteria
* Brain magnetic resonance imaging performed between clinical presentation and treatment
* Cerebrospinal fluid analysis performed between clinical presentation and treatment
* Brain FDG-PET performed between clinical presentation and treatment
* Autoantibodies testing performed between clinical presentation and treatment

Exclusion Criteria:

* Refusal to give consent for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune encephalitis admitted to the recruiting centers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
SPM analysis of brain metabolic pattern | up to 6 months
  Pattern of brain metabolism in patients with autoimmune encephalitis compared with healthy controls and patients with Alzheimer's disease, drawn from validated published databases

SECONDARY OUTCOMES:
Sensitivity of basal ganglia hypermetabolism | up to 6 months
  Sensitivity of basal ganglia hypermetabolism for the diagnosis of autoimmune encephalitis
Diagnostic delay | up to 6 months
  Comparison of diagnostic delay with and without FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: Simone Beretta, MD, PhD, Principal Investigator — University of Milano Bicocca
Locations (6):
- Italy (6):
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Fondazione IRCCS Mondino, Pavia, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Della Brianza
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta", Milan
  - Ospedale San Paolo, Milan

IPD SHARING:
Plan to Share IPD: No